CLINICAL TRIAL: NCT01739218
Title: A Randomized, Open-Label, Phase II Study Assessing the Efficacy and the Safety of Bevacizumab in Neoadjuvant Therapy in Patients With FIGO Stage IIIC/IV Ovarian, Tubal or Peritoneal Adenocarcinoma, Initially Unresectable
Brief Title: A Study of Bevacizumab (Avastin) in Neoadjuvant Therapy in Participants With International Federation of Gynecology and Obstetrics (FIGO) Stage IIIC/IV Ovarian, Tubal, or Peritoneal Cancer, Initially Unresectable
Acronym: ANTHALYA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML28337; 2012-001144-22 (EudraCT Number)
Record Dates: First submitted 2012-11-28; First posted 2012-12-03 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Carboplatin; Paclitaxel; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Carboplatin + Paclitaxel + Bevacizumab (Experimental): Participants will receive 4 cycles of neoadjuvant therapy prior to IDS and 22 cycles of adjuvant therapy before entering long-term follow-up. Each cycle will be 3 weeks in length. Carboplatin and paclitaxel will be administered during Cycles 1 to 8. Bevacizumab will be administered during both the neoadjuvant and the adjuvant treatment periods in Cycles 1 to 26 (no treatment in Cycles 4 and 5).
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Bevacizumab
- Carboplatin + Paclitaxel (Active Comparator): Participants will receive 4 cycles of neoadjuvant therapy prior to IDS and 22 cycles of adjuvant therapy before entering long-term follow-up. Each cycle will be 3 weeks in length. Carboplatin and paclitaxel will be administered during Cycles 1 to 8. Bevacizumab will be administered only during the adjuvant treatment period in Cycles 6 to 26.
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Bevacizumab

INTERVENTIONS:
Drug: Carboplatin — Carboplatin will be administered at a dose calculated according to the Calvert formula ([participant's glomerular filtration rate + 25] multiplied by the target area under the concentration-time curve [AUC] of 5 milligrams per milliliter per minute [mg/mL/min]), as intravenous [IV] infusion over 30-60 minutes [min] every 3 weeks).
Drug: Paclitaxel — Paclitaxel will be administered at a dose of 175 milligrams per meter-squared [mg/m^2] as IV infusion over 3 hours using a rate controlling device every 3 weeks, or at a dose of 80 mg/m^2 as IV infusion over 1 hour using a rate controlling device every week (only during Cycles 5 to 8).
Drug: Bevacizumab — Bevacizumab will be administered at a dose of 15 milligrams per kilogram [mg/kg] as IV infusion over 30-90 min every 3 weeks.
  Other Names: Avastin

SUMMARY:
This randomized, open-label study will evaluate the efficacy and safety of neoadjuvant bevacizumab in participants with initially unresectable, FIGO stage IIIC/IV ovarian, tubal, or peritoneal cancer. Participants will be randomized to receive 8 cycles of carboplatin plus paclitaxel with or without bevacizumab before surgery (interval debulking surgery [IDS]). Surgery will be scheduled 28 days after the last course of neoadjuvant treatment in participants with resectable cancer. Participants with unresectable cancer will go through the follow-up period. All participants will receive bevacizumab for Cycles 6 to 26.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed and documented high-risk FIGO stage IIIC/IV epithelial ovarian carcinoma, fallopian tube carcinoma, or primary peritoneal carcinoma
* Not eligible for primary complete debulking surgery during a laparoscopic procedure as judged by a surgeon experienced in management of ovarian cancer
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2
* Life expectancy greater than or equal to (>/=) 3 months
* Eligible for carboplatin and paclitaxel chemotherapy in accordance with local standards
* Beneficiaries of healthcare coverage under the social security system

Exclusion Criteria:

* Non-epithelial ovarian cancer, ovarian tumor with low malignant potential, mucinous and clear cell ovarian cancer, or carcinosarcoma
* Evidence of abdominal free air not explained by paracentesis or recent surgical procedure
* Previous systemic therapy for ovarian cancer
* Previous exposure to mouse CA-125 antibody
* Current or recent (within 28 days prior to Day 1 of Cycle 1) treatment with another investigational drug or previous participation in this study
* Current or recent (within 10 days prior to first study drug dose) chronic daily treatment with aspirin greater than (>) 325 milligrams (mg) per day
* Planned intraperitoneal cytotoxic chemotherapy
* Inadequate bone marrow, liver, or renal function
* History of myocardial infarction, unstable angina, stroke, or transient ischemic attack within 6 months prior to Day 1 of Cycle 1
* Uncontrolled hypertension
* Clinically significant (active) cardiovascular disease such as New York Heart Association (NYHA) Class II or greater congestive heart failure, or aortic aneurism
* Pre-existing peripheral neuropathy that is Common Toxicity Criteria (CTC) Grade >/=2
* Known hypersensitivity to bevacizumab or its excipients, Chinese hamster ovary cell products or other recombinant humanized antibodies, or to any planned chemotherapy
* Pregnant or lactating females
* History of other clinically active malignancy within 5 years of enrollment, except for tumors with a negligible risk for metastasis or death, such as adequately controlled basal-cell or squamous-cell carcinoma of the skin or carcinoma in situ of the cervix or breast

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2013-02-01 (Actual); Primary Completion 2016-08-17 (Actual); Study Completion 2016-08-17 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Complete Resection After IDS | After IDS (approximately 4 months from randomization)
Percentage of Participants with Different CC Scores After IDS | After IDS (approximately 4 months from randomization)

SECONDARY OUTCOMES:
Percentage of Participants with Objective Response According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) | At IDS (approximately 3 months); at Cycle 26 (approximately 22 months); and at last tumor assessment (up to approximately 38 months)
Percentage of Participants with Response According to Cancer Antigen (CA)-125 Levels | At IDS (approximately 3 months); at Cycle 26 (approximately 22 months); and at last CA-125 assessment (up to approximately 38 months)
Percentage of Participants with RECIST v1.1 Objective Response and CA-125 Response | At Cycle 26 (approximately 22 months) and at last response assessment (up to approximately 38 months)
Percentage of Participants with RECIST v1.1 Objective Response Without CA-125 Response | At Cycle 26 (approximately 22 months) and at last response assessment (up to approximately 38 months)
Percentage of Participants with CA-125 Response Without RECIST v1.1 Objective Response | At Cycle 26 (approximately 22 months) and at last response assessment (up to approximately 38 months)
Number of Participants with Disease Progression or Death From any Cause | From Baseline to disease progression or death due to any cause (up to approximately 38 months)
Progression-Free Survival (PFS) According to RECIST v1.1 | From Baseline to disease progression or death due to any cause (up to approximately 38 months)
Percentage of Participants with Serious Adverse Events (SAEs) and Non-SAEs | SAEs: from randomization up to last assessment (up to approximately 38 months); non-SAEs: from Day 1 up to 28 days after last dose (up to approximately 23 months)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (15):
- France (15):
  - Chu D'Amiens, Amiens
  - HOPITAL JEAN MINJOZ; Oncologie, Besançon
  - Institut Bergonie; Oncologie, Bordeaux
  - Centre Francois Baclesse; Chir Gynecologique, Caen
  - Centre Jean Perrin; Chir Generale Oncologie, Clermont-Ferrand
  - Centre Oscar Lambret; Cancerologie Gynecologique, Lille
  - Institut J Paoli I Calmettes; Chir II, Marseille
  - Centre Val Aurelle Paul Lamarque; Chir A1, Montpellier
  - Centre Antoine Lacassagne; Hopital De Jour A2, Nice
  - Institut Curie; Chir Generale Gyneco Oncologique, Paris
  - Hop Europeen Georges Pompidou; Gynecologie, Paris
  - HOPITAL TENON; Cancerologie Medicale, Paris
  - Centre Rene Huguenin; Chir Generale Oncologique, Saint-Cloud
  - Hopital Rangueil; CHIR Generale Et Gynecologique, Toulouse
  - Institut Gustave Roussy; Departement Chirurgie Generale /Unite Tarn, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gaitskell K, Rogozinska E, Platt S, Chen Y, Abd El Aziz M, Tattersall A, Morrison J. Angiogenesis inhibitors for the treatment of epithelial ovarian cancer. Cochrane Database Syst Rev. 2023 Apr 18;4(4):CD007930. doi: 10.1002/14651858.CD007930.pub3. PMID 37185961